CLINICAL TRIAL: NCT05545813
Title: Impact of Probiotic Supplementation on Cognition and Related Health Outcomes Among Video Gamers: A Randomized, Placebo-Controlled, Double-Blind, Clinical Trial
Brief Title: Impact of Probiotic Supplementation on Cognition and Related Health Outcomes Among Video Gamers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: L-025
Record Dates: First submitted 2022-09-02; First posted 2022-09-19 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-09

CONDITIONS: Stress; Attention Disturbances
Keywords: Attention; Cognition; Acute Stress; Task-switching; Probiotics; HPA-axis
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Participants will be randomized to receive the probiotic formulation for 8 weeks.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Participants will be randomized to receive the placebo formulation for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants will be asked to take 1 capsule (3 billion CFU) daily for 8 weeks in the morning with their first meal.
  Arms: Probiotic
Dietary Supplement: Placebo — Participants will be asked to take 1 capsule daily for 8 weeks in the morning with their first meal.
  Arms: Placebo

SUMMARY:
The primary objective of the current study is to investigate the effect of two probiotic formulations on task-switching following acute stress in healthy, adult action video gamers. It is hypothesized that the participants that consume the probiotic formulations will have improved task-switching performance following acute stress compared to those who consume a placebo.

DETAILED DESCRIPTION:
Participants who are action gamers will be recruited to participate in this randomized, placebo-controlled, 2-arm, parallel trial. Eligible participants will be enrolled in this study for 8 weeks.

The study will consist of 2 laboratory visits: Baseline Visit and Post-Treatment Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 19 to 35 years-old.
2. Have played action video games (i.e., first- and third-person shooter and action role playing games) for a minimum of 5 hours per week over the course of the previous year as assessed by self-report (as per [1])
3. Willingness to continue the same amount of video game playing throughout the duration of the study.
4. Willingness to maintain eating habits throughout the duration of the study.
5. Willingness to discontinue consumption of probiotic supplements and probiotic- fortified products, as well as fiber supplement consumption (e.g., Metamucil, Benefiber, etc.), throughout the duration of the study.
6. Willingness to maintain current physical activity levels throughout the duration of the study.
7. Willing and able to consume a probiotic or placebo supplement for 8 weeks.
8. Willingness to complete questionnaires, records, and diaries associated with the study and to complete all study visits.
9. Able to provide informed consent.

Exclusion Criteria:

1. Use of antidepressants, anti-anxiolytic medication, and/or medication that improves attention, including amphetamines, methylphenidates, dexmethylphenidates, and atomoxetine hydrochloride.
2. Disordered gaming, as per a score above 32 on the Internet Gaming Disorder Scale Short Form (IGDS9-SF; [2]).
3. Head trauma that was diagnosed by a medical professional as a concussion or was associated with a loss of consciousness within the past two years.
4. Currently diagnosed with alcohol use disorder and/or substance use disorder.
5. Diabetes (type I and II), blood/bleeding disorders, liver and/or kidney disorders, unstable cardiovascular diseases, neurological diseases (e.g., Alzheimer's disease, Parkinson's disease, epilepsy), gastrointestinal diseases (e.g., gastric ulcers, Crohn's disease, ulcerative colitis).
6. Presence of unrelated sleep disorders, diagnosis of a mental disorder within the previous year, history of diagnosis of attention-deficit/hyperactivity disorder or attention-deficit disorder
7. Immunodeficiency (immune-compromised and immune-suppressed participants; e.g., AIDS, lymphoma, participants undergoing long-term corticosteroid treatment, chemotherapy and allograft participants).
8. Arthritis pain or other chronic pain.
9. Currently suffering from periodontitis.
10. Pregnancy (as per urine pregnancy test at screening), planning to be pregnant or currently breastfeeding.
11. Females of childbearing potential not using a medically approved method of birth control (e.g. hormonal contraception, intrauterine devices, vasectomy/tubal ligation, barrier methods, double-barrier method) or true abstinence.
12. Milk, soy, and/or yeast allergy.
13. Lactose intolerance.
14. Use of any antibiotic drug within 4 weeks of randomization. Volunteer could be eligible to participate after a 2-week washout period.
15. Current use of probiotics. Volunteer can be eligible after a four (4)-week washout period.
16. Currently enrolled in another clinical trial.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-21 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Change in reaction time | 8 weeks
  The statistical difference in change in reaction time (in milliseconds) from baseline during a computerized task-switching color-word Stroop task following acute stress between the probiotic and placebo groups.

SECONDARY OUTCOMES:
Change in reaction time: acute stress condition | 8 weeks
  The statistical difference in changes in reaction time (in milliseconds) on a computerized incongruent CWST between probiotic and placebo groups following acute stress.
Change in accuracy: acute stress condition | 8 weeks
  The statistical difference in changes in accuracy (proportion correct) on a computerized task-switching CWST and incongruent CWST between probiotic and placebo groups following acute stress.
Change in reaction time: non-stressful condition | 8 weeks
  The statistical difference in changes in reaction time (in milliseconds) on a computerized task-switching and incongruent CWST and a visual search (VS) paradigm, between probiotic and placebo groups in a non-stressful condition.
Change in accuracy: non-stressful condition | 8 weeks
  The statistical difference in changes in accuracy (proportion correct; %false alarms) on a computerized task-switching and an incongruent CWST, a go/no-go paradigm, a visual working memory maintenance paradigm, and a visual working memory complex span task (SYMSPAN) between probiotic and placebo groups in a non-stressful condition.
Change in self-reported cognitive control: non-stressful condition | 8 weeks
  The statistical difference in changes in self-reported cognitive control and cognitive flexibility as per the Cognitive Control and Flexibility Questionnaire (CCFQ) between probiotic and placebo groups in a non-stressful condition.
Changes in oxyhemoglobin concentrations in pre-frontal cortex | 8 weeks
  The statistical difference in changes in concentrations of oxygenated hemoglobin in the prefrontal cortex (PFC) during the task-switching CWST from baseline between the probiotic and placebo groups following acute stress and under non-stress conditions.
Changes in cortisol | 8 weeks
  The statistical difference in changes in the cortisol response to acute stress from baseline, as measured by the area under the curve with respect to increase (AUCi) and with respect to ground (AUCg) between probiotic and placebo groups.
Changes in salivary DHEA-S | 8 weeks
  The statistical difference in salivary DHEA-S from baseline between the probiotic and placebo groups.
Changes in salivary cortisol/DHEA-S ratio | 8 weeks
  The statistical difference in the salivary cortisol/DHEA-S ratio from baseline between the probiotic and placebo groups.
Changes in immune activity markers | 8 weeks
  The statistical difference in changes in salivary levels of proinflammatory cytokines, interleukin-1 beta, and interleukin-6 from baseline between probiotic and placebo groups.
Changes in self-reported levels of depression symptomology | 8 weeks
  The statistical difference in changes in the depression subscale score of the Depression, Anxiety, and Stress Scale Short Form (DASS-21) from baseline between the probiotic and placebo groups.
Changes in self-reported levels of anxiety symptomology | 8 weeks
  The statistical difference in changes in the anxiety subscale score of the Depression, Anxiety, and Stress Scale Short Form (DASS-21) from baseline between the probiotic and placebo groups.
Changes in self-reported levels of perceived stress symptomology | 8 weeks
  The statistical difference in changes in the stress subscale score of the Depression, Anxiety, and Stress Scale Short Form (DASS-21) from baseline between the probiotic and placebo groups.
Changes in self-reported levels of anxiety, depression, and perceived stress symptomology | 8 weeks
  The statistical difference in changes in the total scale score of the Depression, Anxiety, and Stress Scale Short Form (DASS-21) between the probiotic and placebo groups.
Changes in self-reported sleep quality | 8 weeks
  The statistical differences in changes in total Pittsburgh Sleep Quality Index (PSQI) scores between the probiotic and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Perrot, Ph.D., Principal Investigator — Dalhousie University; Heather Neyedli, Ph.D., Principal Investigator — Dalhousie University
Locations (1):
- Cognitive and Motor Performance Lab, Dalplex, Kinesiology Suites, Dalhousie University (Rm. 213), Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
After publications of the results, de-identified data will be shared with qualified researchers and scientists upon reasonable request to the sponsor including a detailed proposal of the intended use of the data, as per the Lallemand Health Solutions Inc. Policy on Clinical Trial Transparency and Data Sharing (available upon request).